CLINICAL TRIAL: NCT00040690
Title: A Clinicopathological Study In Burkitts's And Burkitt-Like Non-Hodgkin's Lymphoma
Brief Title: Combination Chemotherapy in Treating Patients With Burkitt's Lymphoma or Burkitt's Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069374; MRC-LY10; EU-20117
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2007-05

CONDITIONS: Leukemia; Lymphoma
Keywords: untreated adult acute lymphoblastic leukemia; L3 adult acute lymphoblastic leukemia; stage I adult Burkitt lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; contiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult Burkitt lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Burkitt Lymphoma | interventions — Filgrastim; Cyclophosphamide; Cytarabine; Doxorubicin; Etoposide; Ifosfamide; Leucovorin; Methotrexate; Vincristine; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Drug: cyclophosphamide
Drug: cytarabine
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: ifosfamide
Drug: leucovorin calcium
Drug: methotrexate
Drug: vincristine sulfate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients who have Burkitt's lymphoma or Burkitt's leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Describe the morphology, phenotype, and cytogenetics, using fresh tumor tissue (when possible), in patients with Burkitt's or Burkitt-like lymphoma/leukemia treated with the CODOX-M chemotherapy regimen (cyclophosphamide, vincristine, doxorubicin, and methotrexate) alone or alternating with the IVAC chemotherapy regimen (ifosfamide, etoposide, and cytarabine).
* Determine whether cytogenetic and molecular changes are associated with or predictable from the immunophenotype of the tumor cells or patient characteristics (e.g., age).
* Examine the relationship between t(14;18) and bcl-2 expression in patients treated with this regimen.
* Determine whether the presence of specific cytogenetic and molecular changes, in particular the presence of t(14;18) and t(8;14), is associated with an adverse outcome (progression-free and overall survival) in patients treated with this regimen.
* Assess the activity of the alternating CODOX-M/IVAC chemotherapy regimens using a lower dose of methotrexate (compared to the UKLG LY06 trial) in these patients.
* Assess further the activity of these regimens in patients with leukemic Burkitt's lymphoma.
* Modify the chemotherapy doses in these regimens to include older patients who are often excluded from clinical trials.

OUTLINE: This is a multicenter study. Patients with low-risk disease are assigned to group A, while patients with high-risk disease are assigned to group B.

Group A (low-risk group):

* Patients receive 3 courses of the CODOX-M chemotherapy regimen comprising cyclophosphamide IV on days 1-5, vincristine IV on days 1 and 8, doxorubicin IV on day 1, and methotrexate (MTX) IV over 24 hours on day 10. Patients over age 65 receive reduced-dose MTX on day 10. All patients receive leucovorin calcium (CF) IV once at hour 36 after initiation of MTX infusion, once every 3 hours between hours 36-48, and continuing once every 6 hours until blood levels of MTX are safe. Patients also receive filgrastim (G-CSF) subcutaneously (SC) once daily beginning on day 13 and continuing until blood counts recover.
* During all 3 courses of the CODOX-M regimen, patients receive CNS prophylaxis comprising cytarabine (ARA-C) intrathecally (IT) on days 1 and 3, MTX IT on day 15, and oral CF (24 hours after IT MTX) on day 16.

Group B (high-risk group):

* Patients receive the CODOX-M chemotherapy regimen (as above) alternating with the IVAC chemotherapy regimen (as defined below) for a total of 4 courses given in the following sequence: CODOX-M, IVAC, CODOX-M, and IVAC. The IVAC chemotherapy regimen comprises ifosfamide (IFF) IV over 1 hour and etoposide IV over 1 hour on days 1-5 and ARA-C IV over 3 hours on days 1 and 2. Patients over age 65 receive reduced-dose IFF and ARA-C. Patients also receive G-CSF SC once daily beginning on day 7 and continuing until blood counts recover.
* During IVAC, patients without CNS disease receive MTX IT on day 5 and oral CF (24 hours after MTX). Patients with proven CNS disease receive intensified IT therapy throughout the first two courses of CODOX-M/IVAC chemotherapy.

For patients in group B with CNS disease at diagnosis, radiotherapy is only considered in the presence of a cerebral mass documented by CT scan or MRI. Patients in group A or B who develop isolated CNS recurrence (documented by malignant CSF pleocytosis, cranial nerve palsies, or both) at any time after the first course of study therapy receive the same CNS treatment (as above) as patients with proven CNS disease in addition to whole brain irradiation for 3 weeks.

Patients are followed monthly for 4 months, every 2 months for 8 months, every 3 months for 1 year, every 4 months for 1 year, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A minimum of 120 patients (30 with low-risk disease and 90 with high-risk disease) will be accrued for this study within approximately 3-4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of diffuse B-cell lymphoma in a nodal or an extranodal site

  * CD20 and CD79 positive
  * 100% expression of Ki67 (MIB1) in all of the tumor cells OR
* Diagnosis of bone marrow replacement/leukemia comprising mature B-cell lymphoma

  * sIg and CD19 positive
  * CD34 and Tdt negative
* Patients in the low-risk group must meet at least 3 of the following criteria:

  * Normal lactate dehydrogenase (LDH) level
  * WHO performance status 0-1
  * Ann Arbor stage I or II
  * No more than 1 extranodal site (e.g., bone marrow, gastrointestinal tract, or CNS)
* Patients in the high-risk group must meet at least 2 of the following criteria:

  * Raised LDH level
  * WHO performance status 2-4
  * Ann Arbor stage III or IV
  * More than 1 extranodal site

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Performance status:

* See Disease Characteristics

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* See Disease Characteristics

Renal:

* Not specified

Other:

* No mental or physical status that would preclude study
* No other disease or prior malignancy that would preclude study
* HIV negative
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy except 1 course of preinduction chemotherapy (e.g., CHOP [cyclophosphamide, doxorubicin, vincristine, and prednisone] or a related regimen)

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy

Surgery:

* Not specified

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-11; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival

SECONDARY OUTCOMES:
Survival time

CONTACTS AND LOCATIONS:
Overall Officials: Simon Clawson, Study Chair — Medical Research Council
Locations (1):
- Medical Research Council Clinical Trials Unit, London, England, United Kingdom

REFERENCES:
- [Result] Mead GM, Barrans SL, Qian W, Walewski J, Radford JA, Wolf M, Clawson SM, Stenning SP, Yule CL, Jack AS; UK National Cancer Research Institute Lymphoma Clinical Studies Group; Australasian Leukaemia and Lymphoma Group. A prospective clinicopathologic study of dose-modified CODOX-M/IVAC in patients with sporadic Burkitt lymphoma defined using cytogenetic and immunophenotypic criteria (MRC/NCRI LY10 trial). Blood. 2008 Sep 15;112(6):2248-60. doi: 10.1182/blood-2008-03-145128. Epub 2008 Jul 8. PMID 18612102